CLINICAL TRIAL: NCT03811548
Title: A Multicentre, Randomized, Double-blind, Parallel Group, Placebo-controlled Study, to Evaluate the Efficacy and Safety of Janagliflozin (25 mg and 50 mg) as Monotherapy in Chinese Patients Diagnosed With T2DM
Brief Title: Janagliflozin Treat T2DM Monotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5695-DIA-3001
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — janagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Janagliflozin 25mg (Experimental): Each patient will receive 25 mg of Janagliflozin once daily for 52 weeks (24 weeks core period followed by 28 Weeks Extension period)
  Interventions: Drug: Janagliflozin 25mg
- Janagliflozin 50mg (Experimental): Each patient will receive 50 mg of Janagliflozin once daily for 52 weeks (24 weeks core period followed by 28 Weeks Extension period)
  Interventions: Drug: Janagliflozin 50mg
- Placebo/Janagliflozin (Experimental): In the core period, each patient will receive placebo once daily for 24 weeks and will then switch from placebo to 25 mg or 50 mg of Janagliflozin once daily until Week 52.
  Interventions: Drug: Placebo/Janagliflozin

INTERVENTIONS:
Drug: Janagliflozin 25mg — Tablets, Oral, 25 mg, Tablets, Oral, 50 mg
  Other Names: Placebo 50mg
  Arms: Janagliflozin 25mg
Drug: Janagliflozin 50mg — Tablets, Oral, 25 mg, Once daily, 52 weeks
  Other Names: Placebo 25mg
  Arms: Janagliflozin 50mg
Drug: Placebo/Janagliflozin — Tablets, Oral, 25 mg, Once daily, 52 weeks
  Arms: Placebo/Janagliflozin

SUMMARY:
The purpose of this study is to assess the effect of Janagliflozin relative to placebo on glycated hemoglobin (HbA1c) after 24 weeks of treatment, and to assess the efficacy after 52 weeks of treatment, overall safety and Population pharmacokinetics.

DETAILED DESCRIPTION:
A multicentre, randomized, double-blind, parallel group, placebo-controlled study(24 weeks core period followed by 28 Weeks Extension period), to evaluate the efficacy and safety of Janagliflozin (25 mg and 50 mg) compared to placebo in patients diagnosed with T2DM who are not achieving an adequate response from diet and exercise to control their diabetes. Approximately 390 patients with inadequate glycemic control with diet and exercise will receive once-daily double-blind treatment with Janagliflozin 25 mg or 50 mg once daily for 52 weeks, or 24 weeks of double-blind treatment with placebo followed by 28 weeks of single-blind treatment with Janagliflozin 25 mg or 50 mg. During the treatment, if a patient's glycemic level remains high despite treatment with study drug and reinforcement with diet and exercise, the patient will receive treatment with metformin (rescue therapy) consistent with local prescribing information. Study drug will be taken orally once daily.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM (meet the diagnostic criteria for diabetes issued by the World Health Organization in 1999)
* Patients must have a hemoglobin A1c (HbA1c) level ≥7.5% and ≤11% at screening, and ≥7.0% and ≤10.5% at baseline.
* Drug -naïve (never received anti-diabetic medication or did not receive anti-diabetic medication within 8 weeks before screening).
* Body Mass Index: 18.0~35.0 kg/m2 (both inclusive)

Exclusion Criteria:

* History of type 1 diabetes mellitus (T1DM), diabetes caused by pancreatic injury, or secondary diabetes (e.g., diabetes caused by Cushing's syndrome or acromegaly)
* More than 10% change in body weight within the 3 months before screening
* Any laboratory test indicators meet the following standards:

  * fasting plasma glucose ≥ 15 mmol/L
  * aspartate aminotransferase, alanine aminotransferase levels > 3 times the upper limit of normal (ULN); total bilirubin > 1.5 times ULN
  * hemoglobin < 100 g/L
  * eGFR < 60 mL/min/1.73m2
  * fasting triglycerides > 5.64 mmol/L (500 mg/dL)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c From Baseline to Week 24 | Baseline and Week 24
  To examine whether the mean change in HbA1c from baseline to week 24 with Janagliflozin is superiority (superiority margin of 0.5%) to placebo

SECONDARY OUTCOMES:
Change in HbA1c From Baseline to Week 52 | Baseline and Week 52
  To compare the mean change in HbA1c from baseline to week 52 between groups
Percentage of Patients With HbA1c <7% at Week 24 (Core period) and week 52 | Baseline, Week 24 and week 52
  To compare the percentage of patients with HbA1c <7% at week 24 (core period) and week 52 (extension period) between groups
Percentage of Patients With HbA1c <6.5% at Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the percentage of patients with HbA1c <6.5% at week 24 (core period) and Week 52 (extension period) between groups
Change in Fasting Plasma Glucose (FPG) From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in fasting plasma glucose (FPG) from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in 2-hour Post-prandial Glucose From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in 2-hour post-prandial glucose from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Blood Lipids (total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in blood lipids (total cholesterol, triglycerides, high-density lipoprotein cholesterol, and low-density lipoprotein cholesterol) from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Blood Pressure (systolic blood pressure and diastolic blood pressure) From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in blood pressure (systolic blood pressure and diastolic blood pressure) from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Body Weight From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in body weight from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in Fasting C-peptide From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in fasting C-peptide from Baseline to Week 24 (core period) and Week 52 (extension period) between groups.
Change in Insulin Sensitivity From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in insulin sensitivity from Baseline to Week 24 (core period) and Week 52 (extension period) between groups
Change in β-cell Function From Baseline to Week 24 (Core period) and Week 52 (Extension period) | Baseline, Week 24 and Week 52
  To compare the mean change in β-cell function from Baseline to Week 24 (core period) and Week 52 (extension period) between groups.
Percentage of Patients Who Have Received Rescue Therapy at Week 24 (Core period) and Week 52 (Extension period) | Week 24 and Week 52
  To compare the percentage of patients who have received rescue therapy by Week 24 (core period) and Week 52 (extension period) between groups

OTHER OUTCOMES:
Urinary albumin/creatinine ratio (UACR) | From Baseline to Week 52
  To evaluate Urinary albumin/creatinine ratio in different group
Occurrence of adverse events | From Baseline to Week 52
  To evaluate adverse events in different group
Occurrence of hypoglycaemic episodes | From Baseline to Week 52
  To evaluate adverse events in different group
Population pharmacokinetics assessment | Baseline, Week 2, Week4, Week8, Week24
  By compare patients' Minimum Plasma Concentration (on week 2, 4, 8, 24)to eveluate Janagliflozin population pharmacokinetics characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- Linong Ji, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided